CLINICAL TRIAL: NCT05586152
Title: Phase 1/2, Multicenter, Randomized, Double-Masked, Vehicle-Controlled, Multiple Ascending Dose (Part 1) and Optional Dose Expansion (Part 2) Study of INV-102 Ophthalmic Solution in Adult Subjects With Moderate Symptomatic Dry Eye Disease
Brief Title: Study of INV-102 Ophthalmic Solution in Adults With Moderate Symptomatic Dry Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Invirsa, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INV-102-CS-001
Record Dates: First submitted 2022-09-19; First posted 2022-10-19 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye; Keratoconjunctivitis sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- INV-102 0.1% Twice daily (BID) (Experimental): Part 1, Cohort 1: INV-102 ophthalmic solution 0.1% administered twice daily for 2 weeks
  Interventions: Drug: INV-102
- INV-102 0.25% BID (Experimental): Part 1, Cohort 2: INV-102 ophthalmic solution 0.25% administered twice daily for 2 weeks
  Interventions: Drug: INV-102
- INV-102 0.7% BID (Experimental): Part 1, Cohort 3: INV-102 ophthalmic solution 0.7% administered twice daily for 2 weeks
  Interventions: Drug: INV-102
- INV-102 0.7% Three times daily (TID) (Experimental): Part 1, Cohort 4: INV-102 ophthalmic solution 0.7% administered three times daily for 2 weeks
  Interventions: Drug: INV-102
- INV-102 TBD% BID (Experimental): Part 2, Cohort 5: INV-102 ophthalmic solution administered for 2 weeks using a dose based on the results from Part 1, Cohorts 1 to 4
  Interventions: Drug: INV-102
- Vehicle (Placebo Comparator): Part 1 (Cohorts 1-4) and Part 2 (Cohort 5): Vehicle ophthalmic solution administered two or three times daily (dependent on the cohort and the frequency of dosing of INV-102) for 2 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: INV-102 — INV-102 Ophthalmic Solution
  Arms: INV-102 0.1% Twice daily (BID); INV-102 0.25% BID; INV-102 0.7% BID; INV-102 0.7% Three times daily (TID); INV-102 TBD% BID
Drug: Vehicle — Vehicle Ophthalmic Solution
  Arms: Vehicle

SUMMARY:
Phase 1/2, first-in-human, 2-part study to assess topically administered eyedrops of INV-102 during 2-week repeat dosing in subjects with moderate symptomatic dry eye disease. Part 1 will be a Dose Escalation phase across 4 cohorts of subjects to assess safety and tolerability of INV-102, and Part 2 will be an Optional Dose Expansion phase in a fifth cohort of subjects, pending the outcome of Part 1, to assess efficacy of INV-102 in the treatment of moderate symptomatic dry eye disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female subject ≥18 years of age
* Presence of moderate DED in at least one eye

Key Exclusion Criteria:

* Presently using prescription eyedrops, except those used for DED, which must be discontinued 2 weeks prior
* Use of OTC eyedrops except for lubricant eyedrops or artificial tears, within 1 week prior to initiation of study drug dosing
* External eye disease except primary DED
* Systemic disease associated with DED
* History or evidence of ocular infection within the previous 30 days
* History or evidence of ocular herpes simplex or ocular herpes zoster
* Blepharitis or meibomian gland disease requiring the use of either topical or systemic antibiotics within 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Part 1: Characterize the safety profile of INV-102 | Through study completion (Day 22)
  Incidence rate of treatment emergent adverse events (TEAEs)
Part 2: Evaluate the efficacy of INV-102 in an expanded cohort | Day 15
  Change from Baseline to Day 15 in either the Eye Dryness Score -OR- Eye Discomfort Score from the 7-item DED symptom VAS (specific outcome measure for Part 2 will be chosen based on results from Part 1, Cohorts 1 to 4)

SECONDARY OUTCOMES:
Part 2: Evaluate the efficacy of INV-102 using signs and symptoms in a combined outcome score | Day 15
  Change from Baseline to Day 15 in either the Eye Dryness Composite Score -OR- Eye Discomfort Composite Score (outcome measure will be chosen as per Part 2 primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shalwitz, MD, Study Chair — Invirsa, Inc.
Locations (1):
- iuvo BioScience, Rush, New York, United States